CLINICAL TRIAL: NCT01634620
Title: Use of FeNO to Identify Eosinophilic Inflammation in Patients Age 40 Years and Above With Chronic Obstructive Airways Disease
Status: Completed | Type: Observational
Sponsor: Aerocrine AB (Industry)
Responsible Party: Sponsor
Other Study IDs: AER-042
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Chronic Obstructive Airways Disease; Chronic Bronchitis; Chronic Emphysema; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FeNO: Participants with chronic obstructive pulmonary disease (COPD) will have a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit.
  Interventions: Device: NIOX MINO® Instrument (09-1100)

INTERVENTIONS:
Device: NIOX MINO® Instrument (09-1100) — FeNO measurements will be performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011)

SUMMARY:
Objective: To characterize FeNO levels that may be indicative of eosinophilic airway inflammation in patients with chronic obstructive airways disease

Number of participants: Approximately 200 subjects will be enrolled

Reference product: NIOX MINO® Instrument (09-1100)

Performance assessments: Fractional Exhaled Nitric Oxide (FeNO) Measurements will be performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual

Safety assessments: The Investigator is responsible for the detection, reporting, and documentation of events meeting the definition of an Adverse Event (AE) and/or Serious Injuries as provided in this clinical investigation plan from the time that informed consent has been provided and during the study period

Criteria for evaluations: This is an observational, pilot study and there are currently no plans for a formal statistical analysis. Information gained from this study may used to design subsequent studies in patients with chronic obstructive airways disease. Information collected will be summarized in a clinical study report but will not be subject to formal hypothesis testing

DETAILED DESCRIPTION:
INTRODUCTION

Overview:

The measurement of exhaled nitric oxide (FeNO) is the only clinical test for measuring airway inflammation that can be performed consistently and accurately in clinical practice at the point-of-care. Airway inflammation is now recognized as the central mechanism in the pathogenesis of asthma and its symptoms. The measurement of FeNO with the NIOX MINO® device provides a rapid, noninvasive, and inexpensive tool to assess airway inflammation in inflammatory airway diseases such as asthma. The test is easy to perform and requires minimal training for the operator to conduct the test.

Burden of Disease:

Chronic obstructive pulmonary disease (COPD) is a heterogeneous group of diseases characterized by chronic airflow obstruction that interferes with normal breathing . The Centers for Disease Control and Prevention (CDC) reported that in the year 2005, approximately one in 20 deaths in the United States had COPD as the underlying cause.

Role of Exhaled Nitric Oxide (FeNO):

FeNO has evolved as a predictive and prognostic biomarker for airway inflammation. Nitric oxide (NO) gas is produced in the epithelial cells of the bronchial wall as an intrinsic part of the inflammatory process.

COPD can coexist with asthma. However, the exact role of FeNO in patients with established COPD remains to be the defined. While COPD airway inflammation is usually associated with increased neutrophils, some patients with COPD may have features of asthma such as a mixed inflammatory pattern with increased eosinophils. However, many patients have difficulty expectorating sputum and/or can only produce poor quality sputum samples which are not adequate to accurately quantify eosinophilic cells. Since FeNO can be measured easily and reliably, it may be useful in evaluating airway inflammation in COPD and thus predicting steroid responsiveness in COPD.

Intended Use:

NIOX MINO® measures Nitric Oxide (NO) in human breath. Nitric Oxide is frequently increased in inflammatory processes such as asthma. The fractional NO concentration in expired breath (FeNO) can be measured by NIOX MINO® with assurance that such measurements are repeatable and according to guidelines for NO measurement established by the American Thoracic Society.

Rationale for Study:

While there have been a number of preliminary studies on FeNO in COPD, literature defining the role of FeNO in patients with established COPD is minimal. The purpose of the current study, therefore is to characterize FeNO levels that may be indicative of eosinophilic airway inflammation in patients with chronic obstructive airways disease. This data may be useful in determining whether or not FeNO can predict improvement in FEV1 following ICS treatment

CLINICAL INVESTIGATION OBJECTIVES To characterize FeNO levels that may be indicative of eosinophilic airway inflammation in patients with chronic obstructive airways disease.

CLINICAL INVESTIGATION PLAN

This is a pilot, observational, multi-center, single-visit, outpatient study. Subjects meeting all of the Inclusion Criteria and none of the Exclusion Criteria, and who express interest in study participation, will be asked to provide the following documentation and information:

* Informed Consent
* Demographics
* Baseline Characteristics
* FeNO:

  - Subjects will receive training by the study staff on use of the NIOX MINO® device to perform FeNO Measurements
* Spirometry
* Severity of COPD

Subject discharge from the study:

Once all information has been collected and all procedures have been performed, the subject will be discharged from the clinic and their study participation will be complete

Selection of investigation population:

Male and female subjects, age 40 years and above, inclusive, with chronic obstructive pulmonary disease (COPD) including chronic bronchitis and emphysema and/or a mixed diagnosis of asthma/COPD will be recruited. A subject should be withdrawn from the clinical investigation if, in the opinion of the Investigator, it is medically necessary, or if it is the expressed wish of the subject.

Medical device:

The NIOX MINO® was initially cleared by the FDA on March 4, 2008 as a new hand-held device for the measurement of exhaled Nitric Oxide, a marker of eosinophilic airway inflammation. The most recent clearance by the FDA was on September 2, 2010 for Instrument (09-1100), which will be used in this study. NIOX MINO® can be used in children 7-17 years of age and in adults 18 years of age or older in the initial assessment and management of asthma.

The NIOX MINO® is a 10 second test based on exhaled breath measured at a 50 ml/second flow rate. Results are provided at the point of care within 2 minutes after the successful completion of the breath test. The test cannot be influenced by patient effort or variations in the clinician's test technique.

Definitions:

Adverse event: Any incident where the use of a medical device (including in vitro diagnostics) is suspected to have resulted in an adverse outcome in a patient.

Serious Injury means injury or illness that:

* Is life-threatening
* Results in permanent impairment of a body function or permanent damage to a body structure, or
* Necessitates medical or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure.

Malfunction: the failure of a device to meet its performance specifications or otherwise perform as intended.

Caused or contributed: the death or serous injury was or may have been attributed to a medical device, or that the medical device was or may have been a factor in a death or serious injury, including events occurring as a result of:

* Failure
* Malfunction
* Improper or inadequate design
* Manufacture
* Labeling
* User error

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Chronic obstructive pulmonary disease (COPD) including chronic bronchitis and emphysema, and/or a mixed diagnosis of asthma/COPD.

Exclusion Criteria:

* Concurrent Conditions or Disease: Subjects with other chronic obstructive lung diseases including but not limited to cystic fibrosis (CF), bronchiectasis, obliterative bronchiolitis, ciliary dyskinesia, post-viral bronchial hyperresponsive syndrome, vocal cord dysfunction, rhinosinusitis, non-eosinophilic asthma, and reactive airways dysfunction syndrome are excluded. In addition, subjects with pneumothorax, fractured rib(s), or signs of cardiac instability including but not limited to a recent myocardial infarction, unstable angina, unstable vital signs, or acute shortness of breath, chest tightness or chest pain are excluded.
* Study Participation Outside of This Protocol: Subjects currently enrolled in studies of Investigational or non-Investigational Drugs or Medical Devices and/or who participated in these studies within 30 days prior to this study are excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the UNC Hospital Outpatient Pulmonary Function Laboratory in Chapel Hill, NC and approximately 3 to 6 outpatient clinics associated with UNC who meet the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Donohue, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - University of North Carolina Hospitals - Sanford Specialty Clinics, Sanford, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants expressing interest who met inclusion and exclusion criteria were asked to sign written informed consent prior to participation.
Groups:
- FeNO: Participants with chronic obstructive pulmonary disease (COPD) had a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit.
  NIOX MINO® Instrument (09-1100) : FeNO measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011)
Period: Overall Study
Arm/Group | FeNO
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Per-protocol Population
Arm/Group | FeNO
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 80
Region of Enrollment [Number; unit: participants]
  United States | 191
Smoking Status [Number; unit: participants] — At study visit, participants responded to a questionnaire regarding their smoking history. Participants were classified as having never smoked, current smoker, or past smoker.
  participants
    Never Smoked | 9
    Current Smoker | 58
    Past Smoker | 124
Current Medications used for Pulmonary and/or Allergy Conditions [Number; unit: participants] — Provided is a summary of medications taken by >= 5% of participants that are used for pulmonary and/or allergy conditions. The most common medications included short-acting bata-agonist bronchodilators (SABA), inhaled corticosteroid (ICS) and long-acting bata-agonist bronchodilators (LABA) combination products, long-acting antimuscarinic antagonists (LAMA), intranasal corticosteroids, leukotriene receptor antagonists, ICS, and combination SABA/SAMA (short-acting antimuscarinic antagonists)
  participants
    SABA | 160
    ICS/LABA Combination | 144
    LAMA | 133
    Intranasal Corticosteroid | 40
    Leukotriene Receptor Antagonist | 28
    SABA/SAMA | 22
    ICS | 20
    H2-Receptor Antagonist | 18
    Antihistamine | 14
    Histamine H1-Receptor Antagonist | 12
    LABA | 12
    SAMA | 11
    Corticosteroid | 10

OUTCOME MEASURES:

1. Primary Outcome: Spirometry Results: FEV1 (L)
Description: Spirometry values were collected according to American Thoracic Society (ATS) guidelines (ATS, 2005). In the event that spirometry preceded forced exhaled nitric oxide (FeNO) measurements, a wait of not less than 20 minutes was imposed to separate the two procedures. Parameters measured were Forced Expiratory Volume in One Second (FEV1), Forced Vital Capacity (FVC), Forced Expiratory Flow 25-75 (FEF15%-75%), Forced Expiratory Flow 50 (FEF50), and Peak Expiratory Flow (PEF). Spirometry measures the severity of a patient's chronic obstructive pulmonary disease (COPD), with lower scores indicating more severe COPD.
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- FeNO: Participants with chronic obstructive pulmonary disease (COPD) will have a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit.
  NIOX MINO® Instrument (09-1100) : FeNO measurements will be performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011)
Arm/Group | FeNO
Number analyzed (Participants) | 191
Liters | 1.4 (0.67)

2. Primary Outcome: Spirometry Results: FVC (L)
Description: as for outcome 1
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | FeNO
Number analyzed (Participants) | 191
Liters | 2.680 (0.9326)

3. Primary Outcome: Spirometry Results: FEV1 (% Predicted)
Description: as for outcome 1
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Mean (Standard Deviation); unit: Percent Predicted
Arm/Group | FeNO
Number analyzed (Participants) | 191
Percent Predicted | 53.9 (22.11)

4. Primary Outcome: Spirometry Results: FEF50% (L/Sec)
Description: as for outcome 1
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Mean (Standard Deviation); unit: Liters per second
Arm/Group | FeNO
Number analyzed (Participants) | 191
Liters per second | 31.8 (27.78)

5. Primary Outcome: Spirometry Results: FEF25-75 (L/Sec)
Description: as for outcome 1
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Mean (Standard Deviation); unit: Liters per second
Arm/Group | FeNO
Number analyzed (Participants) | 191
Liters per second | 0.759 (0.6898)

6. Primary Outcome: Spirometry Results: PEF (L/Min)
Description: as for outcome 1
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | FeNO
Number analyzed (Participants) | 191
Liters per minute | 244.6 (107.27)

7. Primary Outcome: FeNO Levels by GOLD Stage of Severity
Description: Forced exhaled nitric oxide (FeNO) was measured using a NIOX MINO device. The purpose of this study was to characterize FeNO levels indicative of eosinophilic airway inflammation in patients with chronic obstructive pulmonary disease (COPD). The principal investigator classified subjects into one of four stages of severity using the Global Initiative for Chronic Obstructive Lung Disease (GOLD) severity of COPD stages, with Stage I representing mild COPD severity, Stage II representing moderate COPD severity, Stage III representing severe COPD severity, and Stage IV representing very severe COPD severity (GOLD guidelines, 2012). FeNO levels (in parts per billion or ppb) are summarized for subjects within each category.
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | FeNO
Number analyzed (Participants) | 191
parts per billion (ppb)
  All Subjects (191 subjects) | 15.3 (17.18)
  Stage I (24 subjects) | 13.7 (6.88)
  Stage II (77 subjects) | 18.5 (24.43)
  Stage III (74 subjects) | 13.0 (9.99)
  Stage IV (16 subjects) | 13.0 (8.01)

8. Primary Outcome: FeNO Levels by Inhaled Corticosteroid Use
Description: Forced exhaled nitric oxide (FeNO) was measured using a NIOX MINO device. Reported values are the number of participants with low FeNO (<25 parts per billion or ppb), moderate FeNO (>=25 ppb or <=50 ppb), or high FeNO >50 ppb. Use of Inhaled corticosteroids was measured via a survey during study visit.
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Number; unit: participants
Groups:
- Low FeNO: Participants with chronic obstructive pulmonary disease (COPD) had a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit.
  NIOX MINO® Instrument (09-1100) : FeNO measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011).
  Low FeNo is defined as subjects with FeNo levels <25 parts per billion.
- Moderate FeNO: Participants with chronic obstructive pulmonary disease (COPD) had a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit.
  NIOX MINO® Instrument (09-1100) : FeNO measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011).
  Moderate FeNO is defined as subjects with FeNO levels >=25 parts per billion (ppb) or <=50 ppb.
- High FeNO: Participants with chronic obstructive pulmonary disease (COPD) had a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit.
  NIOX MINO® Instrument (09-1100) : FeNO measurements was performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011).
  High FeNO subjects are defined as subjects with FeNO levels > 50 parts per billion.
Arm/Group | Low FeNO | Moderate FeNO | High FeNO
Number analyzed (Participants) | 170 | 16 | 5
participants
  Use Inhaled Corticosteroids | 143 | 14 | 4
  Do Not Use Inhaled Corticosteroids | 27 | 2 | 1

9. Primary Outcome: FeNO Levels by Smoking Status
Description: Forced exhaled nitric oxide (FeNO) was measured using a NIOX MINO device. Subjects are categorized by low (<25 parts per billion or ppb), moderate (>=25 ppb or <=50 ppb), or high >50 ppb. Subjects were asked if they are a previous or current smoker via a survey during study visit.
Time Frame: Single Visit
Measure: Number; unit: participants
Groups:
- High FeNO: Participants with chronic obstructive pulmonary disease (COPD) had a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit.
  NIOX MINO® Instrument (09-1100) : FeNO measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011).
  High FeNO subjects are defined as subjects with FeNO levels > 50 parts per billion.
Arm/Group | Low FeNO | Moderate FeNO | High FeNO
Number analyzed (Participants) | 170 | 16 | 5
participants
  Previous or Current Smoker | 162 | 15 | 5
  Never Smoked | 8 | 1 | 0

10. Primary Outcome: FeNO Levels by ICD 9 Code Category
Description: Forced exhaled nitric oxide (FeNO) was measured using a NIOX MINO device. Subjects are categorized by low (<25 parts per billion or ppb), moderate (>=25 ppb or <=50 ppb), or high >50 ppb. Based on medical history, subjects were given an Internation Statistical Classification of Diseases and Related Health Problems (ICD) code for concurrent diseases. Of interest, FeNO levels were characterized for subjects coded with chronic obstructive pulmonary disease (COPD) and Asthma, COPD and Emphysema, and then by all other concurrent diseases.
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Number; unit: participants
Arm/Group | Low FeNO | Moderate FeNO | High FeNO
Number analyzed (Participants) | 170 | 16 | 5
participants
  COPD and Asthma | 50 | 7 | 4
  COPD and Emphysema | 46 | 4 | 0
  All other codes | 74 | 5 | 1

11. Primary Outcome: Mean FeNO Levels by ICD 9 Code Category
Description: Forced exhaled nitric oxide (FeNO) was measured using a NIOX MINO device. Based on medical history, subjects were given an International Statistical Classification of Diseases and Related Health Problems (ICD) code for concurrent diseases. Of interest, FeNO levels were characterized for subjects coded with chronic obstructive pulmonary disease (COPD) and Asthma, COPD and Emphysema, and then by all other concurrent diseases.
Time Frame: Single Visit
Population: Per-protocol Population
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | FeNO
Number analyzed (Participants) | 191
parts per billion (ppb)
  COPD and Asthma | 20.5 (27.57)
  COPD and Emphysema | 12.9 (7.40)
  All other codes | 12.9 (8.21)

ADVERSE EVENTS:
Time Frame: Single Visit
Arm/Group | FeNO
Serious Adverse Events (participants affected / at risk) | 2/200
Other Adverse Events (participants affected / at risk) | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FeNO (N=200)
Headache and Chest Discomfort (Cardiac disorders) | 1 (1) — adverse event that was considered serious, severe in severity, not related to performance of the FeNO maneuver, and required no action be taken
Retaining CO2, Jerky Movements (Investigations) | 1 (1) — adverse event that was considered serious, severe in severity, not related to performance of the FeNO maneuver, and required no action be taken

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No